CLINICAL TRIAL: NCT03241316
Title: Antibiotics and Activity Spaces: An Exploratory Study of Behaviour, Marginalisation, and Knowledge Diffusion
Acronym: ESRC
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Mahidol Oxford Tropical Medicine Research Unit (Other); Economic and Social Research Council, United Kingdom (Other); Mae Fah Luang University (Other)
Responsible Party: Sponsor
Other Study IDs: BACN001
Record Dates: First submitted 2017-07-25; First posted 2017-08-07 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Antibiotic Use; Rural Healthcare-seeking Behaviour; Marginalisation (Economic, Social, Spatial)
Keywords: qualitative and survey research

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- district-level representative rural survey: Approximately 4,800 adults in 60 villages across Thailand and Lao PDR to study health and antimicrobial resistance (AMR)-related behaviour in breadth.
  Interventions: Behavioral: Observational study of behaviour
- village-level social network census: Approximately 4,800 adults across 6 villages in rural Thailand and Lao PDR that are exposed to AMR awareness activities to study health behaviour within social networks.
  Interventions: Behavioral: Observational study of behaviour

INTERVENTIONS:
Behavioral: Observational study of behaviour — As a general population survey, our study does not involve a control group. Please note that the investigators do not interview patients; we involve only healthy members of the general public who consider themselves fit to be interviewed.

SUMMARY:
The investigators will conduct two rural surveys in Thailand and Lao PDR to improve the understanding of antibiotic-related health behaviour among the general population. One survey will capture a cross-section of health behaviours that is representative for the rural population in Chiang Rai (Thailand) and Salavan (Lao PDR), the other survey will create a two round village-level panel data set to study the evolution of health behaviours in the context of public engagement activities. The investigators will also collect complementary data about village-level infrastructure through observational check-lists, and collect secondary data on patient load from primary care units catering to their survey villages. As part of the questionnaire testing process, the investigators will conduct (and collect as primary data) cognitive interviews to improve the survey tool, to interpret their data, and to justify their methodological choices.

DETAILED DESCRIPTION:
The investigators will collect two data sets each in Lao PDR and Thailand: the first contains district-level representative health behaviour of approx. 2,400 adults across 30 rural communities per country (4,800 in total; representing rural populations of approx. 1-2 million adults); the second is a complete social network census of approx. 1600 adults each in three rural communities per country (approx. 4,800 in total). Within the sampled villages, the investigators will complete checklists about existing formal and informal healthcare facilities and gather patient load data from primary care units catering to the respective villages. As part of the questionnaire testing process, the investigators will conduct (and collect as primary data) cognitive interviews to improve the survey tool, to interpret our data, and to justify our methodological choices. The investigators will carry out the district-level village survey in one round, and the village-level social network censuses in two rounds. Between the two village social network censuses, the investigators will engage in public engagement activities in the selected villages (focused on antibiotic use) and re-survey all adults in the three villages per country two to three months later.

Objectives:

The primary objective is to improve the understanding of patients' antibiotic-related behaviour to support creative thinking about targeted and unconventional antimicrobial resistance (AMR) interventions in low- and middle-income countries (LMICs).

The investigators strive to achieve this primary objective by informing three research questions in Chiang Rai (Thailand) and Salavan (Lao PDR):

1. What are the manifestations and determinants of problematic antibiotic use in patients' healthcare-seeking pathways?
2. Will people's exposure to antibiotic awareness activities entail changed behaviours that diffuse or dissipate within a network of competing healthcare practices?
3. Which proxy indicators facilitate the detection of problematic antibiotic behaviours across and within communities?

ELIGIBILITY:
Inclusion Criteria:

* Any villager in rural Chiang Rai (Thailand) or Salavan (Lao PDR) who had been sampled to participate in the survey
* Is willing and able to give informed consent for participation in the study
* Is aged 18 years and above

Exclusion Criteria:

* Respondent is not available or able to participate in interview after two attempts to arrange for appointment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Groups included in this study comprise adults (aged 18 years and above) in rural Lao PDR (Salavan) and in rural Thailand (Chiang Rai). As a general population survey, the study does not involve a control group. Please note that the investigators do not interview patients; the investigators involve only healthy members of the general public who consider themselves fit to be interviewed.
  Sampling method:
  1.3-stage stratified random cluster sampling 2.Complete census of all adults among 3 purposively sampled villages per country
Sampling Method: Probability Sample
Enrollment: 5885 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
General population and villagelevel data on antibiotic access and use within individuals' healthcare-seeking pathways | The study is expected to take place from January 2017 to October 2018, with data collection scheduled for November 2017 to April 2018
  To improve the understanding of patients' antibiotic-related behaviour to support creative thinking about targeted and unconventional antimicrobial resistance (AMR) interventions in low- and middle-income countries (LMICs).

SECONDARY OUTCOMES:
Indicators of economic, social, and spatial marginalisation | The study is expected to take place from January 2017 to October 2018, with data collection scheduled for November 2017 to April 2018
  To understand the manifestations and determinants of problematic antibiotic use in patients' healthcare-seeking pathways.
Access to formal and informal medical treatment | The study is expected to take place from January 2017 to October 2018, with data collection scheduled for April 2018.
  To understand the manifestations and determinants of problematic antibiotic use in patients' healthcare-seeking pathways.
Access to prescription and over-the-counter medicines including antibiotics | The study is expected to take place from January 2017 to October 2018, with data collection scheduled for April 2018.
  To understand the manifestations and determinants of problematic antibiotic use in patients' healthcare-seeking pathways.
Degree of technology use during the healthcare seeking process | The study is expected to take place from January 2017 to October 2018, with data collection scheduled for April 2018.
  To understand the manifestations and determinants of problematic antibiotic use in patients' healthcare-seeking pathways.
Awareness about "rational" antibiotic use | The study is expected to take place from January 2017 to October 2018, with data collection scheduled for April 2018.
  To understand the manifestations and determinants of problematic antibiotic use in patients' healthcare-seeking pathways.
Typologies of desirable and undesirable healthcare practices with respect to antibiotic use | The study is expected to take place from January 2017 to October 2018, with data collection scheduled for April 2018.
  To understand whether people's exposure to antibiotic awareness activities entail changed behaviours that diffuse or dissipate within a network of competing healthcare practices.
Social network structures in rural communities | The study is expected to take place from January 2017 to October 2018, with data collection scheduled for April 2018.
  To understand whether people's exposure to antibiotic awareness activities entail changed behaviours that diffuse or dissipate within a network of competing healthcare practices.
Demand fluctuations for healthcare services over time within rural communities | The study is expected to take place from January 2017 to October 2018, with data collection scheduled for April 2018.
  To understand whether people's exposure to antibiotic awareness activities entail changed behaviours that diffuse or dissipate within a network of competing healthcare practices.
Proxy indicators that predict problematic antibiotic use in the general population | The study is expected to take place from January 2017 to October 2018, with data collection scheduled for April 2018.
  To identify less data-intensive indicators to detect problematic contexts of antibiotic use

CONTACTS AND LOCATIONS:
Overall Officials: Marco Haenssgen, Dr., Principal Investigator — Mahidol Oxford Tropical Medicine Unit
Locations (2):
- Lao-Oxford-Mahosot Hospital-Wellcome Trust Research Unit, Vientiane, Laos
- Chiangrai Clinical research Unit, Chiang Rai, Chiangrai, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be de-identified and may be shared with other groups of researchers in accordance with the current MORU Data Sharing Policy provided the respondents consented to data sharing. Specifically, the investigators aim to make their survey data publicly available on the UK Data Service and other local and regional data sharing platforms like the Thai data service in order to enable other researchers the opportunity to study antibiotic-related behaviour in Thailand and Lao PDR.
Supporting Information: Study Protocol, ICF
Time Frame: Data access on the UK Data Service will be free and without a case-by-case assessment, provided repository users agree to the terms and conditions of the UK Data Service and to cite the data sources in all publications emerging from the data, using suggested citations. Data preparation and documentation process will commence in May 2018; deposition will take place within three months of project completion. The data sets will also be utilised as training resources in the context of global health education and social network analysis
Access Criteria: Direct access will be granted to authorised representatives from the sponsor or host institution for monitoring and/or audit of the study to ensure compliance with regulations. Following data entry and validation, we will deposit the de-identified quantitative survey data with the UK Data Service for open access. Data access will be free and without a case-by-case assessment, provided repository users agree to the terms and conditions of the UK Data Service and to cite the data sources in all publications emerging from the data, using suggested citations (see Section 10.6 on Data Sharing for further details). The qualitative data from the cognitive interviews will not be made open access or shared with other researchers.
URL: http://www.surveycto.com/index.html

REFERENCES:
- [Derived] Haenssgen MJ, Charoenboon N, Xayavong T, Althaus T. Precarity and clinical determinants of healthcare-seeking behaviour and antibiotic use in rural Laos and Thailand. BMJ Glob Health. 2020 Dec;5(12):e003779. doi: 10.1136/bmjgh-2020-003779. PMID 33298471
- [Derived] Haenssgen MJ, Charoenboon N, Zanello G, Mayxay M, Reed-Tsochas F, Lubell Y, Wertheim H, Lienert J, Xayavong T, Khine Zaw Y, Thepkhamkong A, Sithongdeng N, Khamsoukthavong N, Phanthavong C, Boualaiseng S, Vongsavang S, Wibunjak K, Chai-In P, Thavethanutthanawin P, Althaus T, Greer RC, Nedsuwan S, Wangrangsimakul T, Limmathurotsakul D, Elliott E, Ariana P. Antibiotic knowledge, attitudes and practices: new insights from cross-sectional rural health behaviour surveys in low-income and middle-income South-East Asia. BMJ Open. 2019 Aug 20;9(8):e028224. doi: 10.1136/bmjopen-2018-028224. PMID 31434769
- [Derived] Haenssgen MJ, Charoenboon N, Zanello G, Mayxay M, Reed-Tsochas F, Jones COH, Kosaikanont R, Praphattong P, Manohan P, Lubell Y, Newton PN, Keomany S, Wertheim HFL, Lienert J, Xayavong T, Warapikuptanun P, Khine Zaw Y, U-Thong P, Benjaroon P, Sangkham N, Wibunjak K, Chai-In P, Chailert S, Thavethanutthanawin P, Promsutt K, Thepkhamkong A, Sithongdeng N, Keovilayvanh M, Khamsoukthavong N, Phanthasomchit P, Phanthavong C, Boualaiseng S, Vongsavang S, Greer RC, Althaus T, Nedsuwan S, Intralawan D, Wangrangsimakul T, Limmathurotsakul D, Ariana P. Antibiotics and activity spaces: protocol of an exploratory study of behaviour, marginalisation and knowledge diffusion. BMJ Glob Health. 2018 Mar 28;3(2):e000621. doi: 10.1136/bmjgh-2017-000621. eCollection 2018. PMID 29629190